CLINICAL TRIAL: NCT06193460
Title: Evaluation of the Anti-anaesthetic Effects of Low-Level Laser Therapy on Children's Soft Tissue Randomized Clinical Trial
Brief Title: Evaluation of the Anti-anaesthetic Effects of Low-Level Laser Therapy on Children's Soft Tissue
Acronym: laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Alaa M Eldehna, lecturer of paediatric dentistry, Al-Azhar University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: ODHOD-101-1Q
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Local Anesthetic Complication
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Group I (20 teeth): the anaesthesia will be reversed by the photobiomodulation mode of diode laser therapy (low-level laser therapy).
  Group II (controlled group) :( 20 teeth) anaesthesia will be withdraw without intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser group (Experimental): The anaesthesia will be reversed by the photobiomodulation mode of the diode laser (low-level laser therapy).
  Interventions: Device: low-level laser therapy
- control group (No Intervention): The anesthesia will be withdrawn without intervention.

INTERVENTIONS:
Device: low-level laser therapy — photobiomodulation mode of diode laser (low-level laser therapy).
  Arms: laser group

SUMMARY:
Evaluate the effect of the photobiomodulation mode of the diode laser on the anaesthetic area and find the best parameter that would accelerate the withdrawal of anaesthesia.

DETAILED DESCRIPTION:
A randomized clinical trial will be performed at the Pedodontics Out Paediatric Clinic at the Facility of Dental Medical for girls. Al Azhar University has twenty patients with upper or lower first primary molars on the right and left sides that need to be treated. Using the split-mouth technique, the mouth will be split in two halves. The first half represents the first group, and the second half represents the second group.

Group I (20 teeth): the anaesthesia will be reversed by the photobiomodulation mode of diode laser (low-level laser therapy).

Group II (controlled group): 20 teeth of anesthesia will be withdrawn without intervention.

To avoid bias in the 2nd group, the laser will be applied on this side, but in turned-off mode. The type of anaesthesia that will be evaluated is articine hydrochloride 4% with 1:200 epinephrine (vasoconstrictor).

ELIGIBILITY:
Inclusion Criteria:

Parents have to complete the written consent form. Patient who behaved well. Children aged from 6 to 12 years can evaluate soft tissue anaesthesia. Patients that require treatment with bilateral upper or lower first primary molar infiltration under anaesthesia.

Exclusion Criteria:

Patients who are mentally disordered or hand-capped. uncooperative patients.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Outcomes measuring the duration (in minutes) of anaesthesia withdrawal after laser application | after application of laser immediately and continue each 15 minutes till complete withdrawal of anaesthesia
  1. Return the normal sensation to the lip.
  2. Being able to smile, drink, and talk normally.
  3. Return of pain sensation that result from the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
A randomized clinical trial will be performed at the Pedodontics Out Paediatric Clinic at the Facility of Dental Medical for girls. Al Azhar University has twenty patients with upper or lower first primary molars on the right and left sides that need to be treated. Using the split-mouth technique, the mouth will be split in two halves. The first half represents the first group, and the second half represents the second group.
  Laser Group: (20 teeth) The anaesthesia will be reversed by the photobiomodulation mode of the diode laser (low-level laser therapy).
  Controlled Group: (20 teeth) anaesthesia will be withdrawn without intervention.